CLINICAL TRIAL: NCT04106349
Title: REPLICA: Real Patient Life Treatment With Cabozantinib in Monotherapy or in Combination With Nivolumab in Patients With Advanced or Metastatic RCC: a Descriptive and Prospective Non Interventional Study.
Brief Title: Observational Real-life Study of Cabozantinib in Monotherapy or in Combination With Nivolumab in Advanced Renal Cell Carcinoma (RCC)
Acronym: REPLICA
Status: Active, not recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-BE-60000-047
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1st line
- 2nd line
- later lines

SUMMARY:
The purpose of this study is to describe the real-life use of Cabometyx® in monotherapy or in combination with nivolumab in Belgium in patients with advanced or metastatic Renal Cell Carcinoma (1st, 2nd and later lines of treatment)

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years and older
* Patients scheduled to receive Cabometyx® in monotherapy or in combination with nivolumabfor advanced or metastatic renal cell carcinoma
* Decision to treat patients with Cabometyx® in monotherapy or in combination with nivolumab has to be taken prior to and independent from participation in the clinical study
* Provision of written informed consent

Exclusion Criteria:

* Participation in another interventional clinical study at the same time
* Previous participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced or metastatic renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment line | Baseline
  Treatment line will be assessed at baseline. It is a percentage of patients receiving cabozantinib as 1st, 2nd or later lines of treatment or cabozantinib in monotherapy or in combination with nivolumab as 1st line of treatment.
Dose reductions and reasons | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
  Number of dose reductions and reason
Treatment interruptions and reason | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
  Number of treatment interruptions and reason
Treatment discontinuations and reason | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
  Number of patients with permanent discontinuation and reason
Alternative dose schedule | From baseline until the end of study up to 9 months
  Number of patients with schedules other than 1 pill at fixed dose/day for the total treatment period
Mean number of any dose modification | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
Median number of any dose modification | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
Median time to any first dose modification | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
Median time to end of treatment | From baseline until the end of study up to 9 months
Duration of treatment exposure | From baseline until the end of study up to 9 months
Dose prescribed at initiation | Baseline
  Number of patients with dose of 60 mg/day, 40 mg/day or 20 mg/day at baseline
Average daily dose | From baseline until the end of study up to 9 months
  Estimation of average daily dose received by subject during the treatment exposure

SECONDARY OUTCOMES:
Change in Quality of Life score | From baseline up to 6 to 8 weeks after cabozantinib initiation and within 10 days of cabozantinib stop
  Changes in quality of life data by comparing changes in scores on Using the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Kidney Symptom Index-19 (NFKSI-19). It describes the severity, interference, and frequency rates.
Progression Free Survival (PFS) | From baseline until the end of study up to 9 months
  Radiological progression using RECIST 1.1 or investigator assessed or according to local standard of care or death; PFS evaluated at least every 12 weeks under treatment with cabozantinib
Objective Response Rate | From baseline until the end of study up to 9 months
  Percent of patients with partial and complete response during the treatment with cabozantinib
Disease Control Rate | From baseline until the end of study up to 9 months
  Percent of patients with stable disease, partial and complete response during the treatment with cabozantinib

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (20):
- Belgium (20):
  - Onze-Lieve-vrouw Ziekenhuis Aalst, Aalst
  - Imeldaziekenhuis, Bonheiden
  - Clinique Saint-Luc Bouge, Bouge
  - AZ Sint-Jan Brugge, Bruges
  - AZ Sint-Lucas, Bruges
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg Genk, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Hôpital de Jolimont, La Louvière
  - CHC MontLegia, Liège
  - CHR Citadelle Liège, Liège
  - CHU Liège / Sart-Tilman, Liège
  - Hôpital Ambroise-Paré Mons, Mons
  - CHU Charleroi - site André Vésale, Montigny-le-Tilleul
  - Clinique Saint-Pierre, Ottignies
  - AZ Delta, Roeselare
  - AZ Glorieux, Ronse
  - CHWAPI, Tournai
  - AZ Turnhout, Turnhout
  - CHR Verviers, Verviers

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/